CLINICAL TRIAL: NCT05456230
Title: Comparison of Postoperative Delirium in Elders Anaesthetised With Midazolam and Without Midazolam During Non-cardiac Surgery
Brief Title: Comparison of Postoperative Delirium in Elders Anaesthetised With Midazolam and Without Midazolam
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); China-Japan Friendship Hospital (Other); Fudan University (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Taihe Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-POD-001
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Midazolam; Benzodiazepines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midazolam: Midazolam as a premedication was given as the patient is taken to the operating room and typically within 15 minutes of anesthetic induction.
  Interventions: Drug: Midazolam
- Non-Midazolam: Midazolam was not given during the operation.

INTERVENTIONS:
Drug: Midazolam — Midazolam as a premedication was given as the patient is taken to the operating room and typically within 15 minutes of anesthetic induction.
  Other Names: benzodiazepines
  Groups: Midazolam

SUMMARY:
This research project is an observational cohort study by prospective chart review of patients that underwent surgery in multi-centers, China, in the years 2020-2022. The purpose of this study is to compare the occurrence of postoperative delirium With Midazolam and Without Midazolam During Non-cardiac Surgery in Elders.

DETAILED DESCRIPTION:
Post operative delirium will be diagnosed using the 3D- CAM(Confusion Assessment Method) which tests for four features with a series of questions. The features include 1) acute onset and fluctuating course,2) inattention,3) disorganized thinking and 4) altered level of consciousness. Diagnosis of delirium is made if features 1 and 2 and either 3 or 4 are present.

The demographic data of the patients,type and site of surgery will be noted. Preoperative hemoglobin, serum electrolytes and blood urea will be recorded. The intraoperative factors like duration of surgery and anaesthesia,use of intravenous fluids ,blood loss, number blood units transfused and opioid use will be studied at the time of surgery. The time to emergence and extubation following the completion of surgery will be noted.

The postoperative factors like postoperative pain, nausea and vomiting, fever,hemoglobin,serum electrolytes and blood urea will be noted.

Preoperative and postoperative pain will be assessed using the numerical rating score on a scale of one to ten.

The association of various preoperative,intraoperative and postoperative factors with POD will be determined.

ELIGIBILITY:
Inclusion Criteria:

Geriatric surgical patients ≥65 years old Underwent elective non-cardiac surgery

Exclusion Criteria:

History of neuropsychiatric diseases including delirium, mental disorders, Parkinson, dementia, etc.; The operation was cancelled due to various reasons after the patient was enrolled; severe liver disease; severe renal dysfunction defined as either having creatinine clearance < 30 ml/min or being dialysis-dependent; Patients who undergo second operation in a short period; Refused to participate in the study.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 11927 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Day 1 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of postoperative delirium | Day 2 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of postoperative delirium | Day 3 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of postoperative delirium | Day 4 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of postoperative delirium | Day 5 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily
Incidence of postoperative delirium | Day 7 postoperatively
  Occurrence of delirium on any postoperative day, as assessed using the 3D-CAM or CAM-ICU daily

SECONDARY OUTCOMES:
the incidence of survival rate | 1 year
  collection of clinical data in the medical record and follow-up update

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No